CLINICAL TRIAL: NCT07327164
Title: Precision Medicine in Neurocutaneous Syndromes: Genotype-Guided Risk Stratification and Targeted Therapy Outcomes in a 20-Year Multicenter Cohort From Western China
Brief Title: Precision Medicine for Neurocutaneous Syndromes in Western China
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other); Xinqiao Hospital, Amry Medical University (Unknown)
Responsible Party: Principal Investigator, Zhigang Lan, Professor, West China Hospital
Other Study IDs: WestChinaH-HX-2025-08
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-01

CONDITIONS: Neurocutaneous Syndromes; Neurofibromatosis Type 1 (NF1); Tuberous Sclerosis Complex (TSC); Sturge-Weber Syndrome (SWS); Von Hippel-Lindau Disease
Keywords: Precision Medicine; Targeted Therapy; Western China; cost-effectiveness
MeSH Terms: conditions — Neurocutaneous Syndromes; Neurofibromatosis 1; Tuberous Sclerosis; Sturge-Weber Syndrome; von Hippel-Lindau Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multidisciplinary Care Group: patients referred to or enrolled in a structured telemedicine-supported multidisciplinary clinic, which included scheduled virtual visits via WeChat Video or DingTalk with neurologists, genetic counselors, and specialty nurses. Real-time interpretation was available for ethnic minority patients.
- Standard In-Person Care (SIC) Group: Patients managed through conventional outpatient visits without structured telemedicine support.

SUMMARY:
The goal of this observational study (retrospective multicenter cohort study) is to learn if precision medicine approaches-including genetic testing, targeted drugs, and coordinated care from multiple specialists-can improve health outcomes and lower medical costs for people with neurocutaneous syndromes (NCS) in Western China, where healthcare resources are limited. NCS includes four main conditions: neurofibromatosis type 1 (NF1), tuberous sclerosis complex (TSC), Sturge-Weber syndrome (SWS), and von Hippel-Lindau disease (VHL). The main questions it aims to answer are:

* Do genetic testing and targeted drugs help people with NCS live longer without disease getting worse?
* Do these approaches better control seizures (for TSC and SWS) and shrink tumors (for NF1 and VHL)?
* Do they reduce the total cost of medical care?

Researchers will compare two groups to see the effects: participants who received precision medicine (genetic testing + targeted drugs + multidisciplinary care) versus those who received standard, uncoordinated care.

Participants will:

* Undergo genetic testing to identify specific gene changes linked to their NCS
* Receive targeted drugs (e.g., mTOR inhibitors for TSC, MEK inhibitors for NF1) if eligible
* Attend regular checkups, imaging scans (like MRI), and follow-up visits for an average of 11.4 years
* For those in the multidisciplinary care group, receive coordinated care from neurologists, geneticists, surgeons, and other specialists (with remote telemedicine visits for those living far from hospitals)

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of one of the following neurocutaneous syndromes: Neurofibromatosis Type 1 (NF1) Tuberous Sclerosis Complex (TSC) Sturge-Weber Syndrome (SWS) Von Hippel-Lindau Disease (VHL) (Diagnosis established by established clinical criteria [e.g., NIH criteria for NF1, International TSC Consensus Criteria] or confirmed pathogenic genetic variant)

* Age between 0 and 65 years at the time of initial evaluation.
* Follow-up duration of at least 12 months at one of the participating tertiary medical centers in Western China:

West China Hospital, Sichuan University (Chengdu) Xinqiao Hospital, Army Medical University (Chongqing) The First Affiliated Hospital of Xi'an Jiaotong University (Xi'an)

*Availability of complete baseline clinical data, including: Demographic information Diagnostic workup Initial symptom profile Treatment history (if any)

Exclusion Criteria:

* Incomplete medical records- Key clinical, imaging, or genetic data missing, preventing reliable diagnosis or outcome assessment.
* Follow-up duration less than 12 months- Patients lost to follow-up or with insufficient longitudinal data to evaluate clinical outcomes.
* Diagnostic uncertainty- Cases that did not meet established clinical or genetic diagnostic criteria for NF1, TSC, SWS, or VHL (e.g., atypical presentations without molecular confirmation).
* Age > 65 years at initial evaluation- Although rare in neurocutaneous syndromes, patients older than 65 were excluded to maintain cohort relevance to typical disease onset and progression patterns.
* Participation in another interventional trial during the study period (if applicable)

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included 1200 patients with neurocutaneous syndromes (NF1, TSC, SWS, or VHL) from three tertiary hospitals in Western China, recruited between 2015 and 2023. Participants were aged 0-65 years (median age at diagnosis: 8.2 years), with 69.3% under 18 years old and a slight male predominance (53.6%). All had confirmed diagnoses and at least 12 months of follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 12 months
  Proportion of patients from diagnosis to disease progression, malignant transformation, or death
Seizure control | 12 months
  Engel class I/II refers to the **Engel Epilepsy Surgery Outcome Scale**, a widely used classification system for assessing seizure control after epilepsy surgery. It categorizes patients into four classes based on postoperative seizure frequency:
  1. **Engel Class I**: **Seizure-free** or **auras only** (no disabling seizures).
  2. **Engel Class II**: **Rare disabling seizures** (≤3 seizure days per year). Higher Engel class (I > II > III > IV) indicates better seizure control.
Tumor response | 12 months
  volumetric tumor reduction measured with preoperative tumor volume
Quality of life: SF-36 Score | 12 months
  SF-36 (Short-Form 36) is a 36-item patient-reported survey that measures generic health-related quality of life across eight domains and two summary components. Each domain is scored 0-100, where 0 = maximum disability and 100 = no disability; therefore, **higher values always indicate better health**.
  Domain structure and score range
  1. **Physical functioning (PF)** - 0-100
  2. **Role-physical (RP)** - 0-100
  3. **Bodily pain (BP)** - 0-100 (higher = less pain)
  4. **General health (GH)** - 0-100
  5. **Vitality (VT)** - 0-100
  6. **Social functioning (SF)** - 0-100
  7. **Role-emotional (RE)** - 0-100
  8. **Mental health (MH)** - 0-100

SECONDARY OUTCOMES:
Overall survival Rate | 12 months
  the overall survivial rate in the whole cohort
treatment costs | 12 Months
  the amount of money(Chinese Yuan, ¥) in volved in the medical costs and transportation costs

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol